CLINICAL TRIAL: NCT04037384
Title: Alternative Home Training Possibilities for Glaucoma Patients
Brief Title: Training of Eye Movements in Glaucoma
Acronym: EyeYoga
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Magdeburg (Other)
Responsible Party: Principal Investigator, Bernhard A. Sabel, Head of Institute, Professor, University of Magdeburg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UMagdeburg
Record Dates: First submitted 2019-07-03; First posted 2019-07-30 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Glaucoma; Eye Yoga
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eye Yoga group (Active Comparator): Eye yoga exercises
  Interventions: Behavioral: Passive Reading
- Reading Group (Placebo Comparator): Passive reading
  Interventions: Behavioral: Eye yoga

INTERVENTIONS:
Behavioral: Eye yoga — Eye yoga exercises at home given by a trained instructor
  Arms: Reading Group
Behavioral: Passive Reading — Passive reading at home
  Arms: Eye Yoga group

SUMMARY:
The aim of the trial is to investigate the possibilities of improving visual impairments with eye training exercises (eye-yoga) in a total of 40 patients with glaucoma who have not previously been treated within a similar training program. 20 patients will be instructed how to do eye yoga to be performed dails for 4 weeks (max 30 min/day). As a control group of 20 patients will be instructed to read for 30 min/day for 4 weeks.

The following outcome measures will be investigated: High Resolution Perimetry, Humphrey Perimetry, Visual Acuity Test, Contrast Sensitivity Test, Microsaccades measurements, Intraocular Pressure Measurement, Electroencephalogram (EEG), Blood Pressure and Pulse Measurement and Dynamic Vessel Analysis (DVA - the blood supply in the eye (especially vascular dysregulation) .

Furthermore, factors that could influence response variability and the effectiveness of treatment will be analysed: (i) the role of mental stress (or stress resilience) and (ii) the influence of personality traits and quality of life.

The study is intended to further validate this home training program (eye yoga) for the treatment of visual impairment in glaucoma.

DETAILED DESCRIPTION:
The aim of eye yoga is to improve microsaccade impairments in patient with primary open angle glaucoma. We will study how this affects visual performance and the physiology of the eye and brain

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of glaucoma
* residual vision
* the duration of the disease must be at least 6 months old
* the visual field defect must be stable

Exclusion Criteria:

* autoimmune diseases in the acute stage
* neurological and mental diseases
* diabetic retinopathy
* addictions
* hypertension (maximum 160/100 mmHg)
* retinitis pigmentosa-
* pathological nystagmus
* non-distant tumors or recurrent tumors
* photosensitivity
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Visual field size determined by perimetry measurements | 4 weeks
  Changes of the visual field's size, evaluated by static perimetry and high resolution perimetry measurements
Microsaccade measurements | 4 weeks
  Changes in the deviation of eye movements when visual targets are followed, using a computerized test

SECONDARY OUTCOMES:
Blood circulation in the eye | 4 weeks
  Changes of the diameter of blood vessels in the eye, measured by vessel analysis
EEG connectivities | 4 weeks
  Changes in alpha power using EEG recording (128 channels)

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard A Sabel, PhD, Principal Investigator — University of Magdeburg
Locations (2):
- Germany (2):
  - Inst. of Medical Psychology, Univ. of Magdeburg, Magdeburg
  - Institute of Medical Psychology, Magdeburg

IPD SHARING:
Plan to Share IPD: Yes
The results will be available without restriction
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the results are published, unlimited duration
Access Criteria: Contact to the principal investigator

REFERENCES:
- [Background] Dada T, Mittal D, Mohanty K, Faiq MA, Bhat MA, Yadav RK, Sihota R, Sidhu T, Velpandian T, Kalaivani M, Pandey RM, Gao Y, Sabel BA, Dada R. Mindfulness Meditation Reduces Intraocular Pressure, Lowers Stress Biomarkers and Modulates Gene Expression in Glaucoma: A Randomized Controlled Trial. J Glaucoma. 2018 Dec;27(12):1061-1067. doi: 10.1097/IJG.0000000000001088. PMID 30256277
- [Background] Sabel BA, Flammer J, Merabet LB. Residual vision activation and the brain-eye-vascular triad: Dysregulation, plasticity and restoration in low vision and blindness - a review. Restor Neurol Neurosci. 2018;36(6):767-791. doi: 10.3233/RNN-180880. PMID 30412515
- [Derived] Zhou W, Sabel BA. Vascular dysregulation in glaucoma: retinal vasoconstriction and normal neurovascular coupling in altitudinal visual field defects. EPMA J. 2023 Feb 16;14(1):87-99. doi: 10.1007/s13167-023-00316-6. eCollection 2023 Mar. PMID 36866155